CLINICAL TRIAL: NCT06435624
Title: Effectiveness of Intelligent Rehabilitation Robot Training System Combined With Repetitive Facilitative Exercise on Upper Limb Motor Function After Stroke: a Randomized Control Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Mingzhou Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jingzhi Zhang, technician, Nanjing Mingzhou Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NJKF202401001
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IRAT group (Experimental): The Intelligent robotic-assisted training (IRAT) group received a 30 minute RFE intervention and a 30 minute IRAT intervention.
  Interventions: Device: intelligent robotic-assisted training; Other: repetitive facilitative exercise
- RFE group (Active Comparator): The Repetitive facilitative exercise (RFE) group received a 60 minute RFE intervention.
  Interventions: Other: repetitive facilitative exercise
- CT group (Active Comparator): The Conventional therapy (CT) group received a 60 minute conventional rehabilitation intervention.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Device: intelligent robotic-assisted training — Using an intelligent robotic-assisted training (IRAT) system to simulate a real work environment, providing functional oriented treatment for stroke patients and improving upper limb motor function.
  The instrument used is the Burt upper limb robot training system produced by Estun Medical Co., Ltd.
  Arms: IRAT group
Other: repetitive facilitative exercise — Repetitive facilitative exercise (RFE) is a new technology that combines multiple sensory stimuli and achieves facilitation and reinforcement of the reconstruction of paralyzed neural pathways through repeated and extensive directional exercise.
  Arms: IRAT group; RFE group
Other: conventional therapy — Basic training, including passive joint movement and activities of daily living exercise.
  Arms: CT group

SUMMARY:
The goal of this clinical trial is to learn if intelligent rehabilitation robot training system combined with repetitive facilitative exercise (RFE) work to treat stroke in adults. The main questions it aims to answer are:

Does drug intelligent rehabilitation robot training system combined with RFE improve the upper limb motor function of participants? Can the combination of intelligent rehabilitation robot training system and RFE achieve better effects?

Researchers will compare 3 groups (RFE, intelligent rehabilitation robot training system under RFE, and conventional therapy) to see if intelligent rehabilitation robot training system and RFE works to treat stroke.

Participants will:

Receive treatment for 4 weeks Receive scale and instrument testing before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* patients (18 to 74 years old) who suffered a first or second unilateral stroke
* chronic stroke (over 6 months from the onset)
* obvious upper limb movement disorders (FMA-UE scores from 25 to 42)
* ability to understand and follow simple directions

Exclusion Criteria:

* pregnant or lactating
* upper extremity contracture, pain, or trauma
* perceptual, apraxic, or cognitive deficits that lead to inability to follow verbal instructions
* unable to maintain sitting posture
* cerebellar lesion
* clinically unstable medical disorders
* inability to provide informed consent

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Mingzhou Rehabilitation Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhang JZ, Chen J, Liu XL, Yan LB, Xu SM. Effectiveness of intelligent robotic-assisted training system combined with repetitive facilitative exercise on upper limb motor function after stroke: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Jul 3;17(1):178. doi: 10.1186/s13102-025-01234-y. PMID 40611355

RESULTS

PARTICIPANT FLOW:
Groups:
- IRAT Group: The Intelligent robotic-assisted training (IRAT) group received a 30 minute RFE intervention and a 30 minute IRAT intervention.
  intelligent robotic-assisted training: Using an intelligent robotic-assisted training (IRAT) system to simulate a real work environment, providing functional oriented treatment for stroke patients and improving upper limb motor function.
  The instrument used is the Burt upper limb robot training system produced by Estun Medical Co., Ltd.
  repetitive facilitative exercise: Repetitive facilitative exercise (RFE) is a new technology that combines multiple sensory stimuli and achieves facilitation and reinforcement of the reconstruction of paralyzed neural pathways through repeated and extensive directional exercise.
Period: Overall Study
Arm/Group | IRAT Group | RFE Group | CT Group
Started | 27 | 27 | 27
Completed | 25 | 26 | 25
Not Completed | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IRAT Group | RFE Group | CT Group | Total
Number analyzed (Participants) | 25 | 26 | 25 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (12.3) | 46.8 (11.7) | 50.3 (14.0) | 49.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 15 | 16 | 16 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 25 | 26 | 25 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 25 | 26 | 25 | 76
Affected side, left/right [Number; unit: participants]
  left | 12 | 12 | 14 | 38
  right | 13 | 14 | 11 | 38
Time from stroke, days [Mean (Standard Deviation); unit: days] | 256.2 (60.1) | 254.7 (46.0) | 270.1 (55.8) | 260.3 (53.9)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment for Upper Extremity (FMA-UE)
Description: The FMA-UE consists of 33 items across nine components, including reflex action, synergy, and coordination, with a maximum score of 66 points. Each items is scored from 0 (no ability) to 2 (full ability), with higher scores indicating better upper limb motor function.
Time Frame: From enrollment to the end of treatment at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IRAT Group | RFE Group | CT Group
Number analyzed (Participants) | 25 | 26 | 25
score on a scale
  baseline | 34.4 (3.5) | 34.9 (3.8) | 35.8 (3.9)
  4 weeks | 49.0 (3.3) | 44.2 (3.6) | 38.8 (3.8)

2. Primary Outcome: Active Participation Proportion
Description: Active Participation Proportion (APP) is measured using the benchmark evaluation system within the intelligent rehabilitation robot training system. The robotic arm's mechanical sensor continuously detects the force exerted by the patient during the test game and quantifies APP as the ratio of the patient's applied force to the total force required to complete the task (%). A higher APP indicates greater voluntary effort in movement execution. Since the test game difficulty is fixed, APP increases as the patient's motor ability improves.
Time Frame: From enrollment to the end of treatment at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of active participation
Arm/Group | IRAT Group | RFE Group | CT Group
Number analyzed (Participants) | 25 | 26 | 25
percentage of active participation
  baseline | 61.7 (4.8) | 104.0 (7.9) | 60.8 (6.1)
  4 weeks | 80.4 (5.3) | 61.6 (2.8) | 60.9 (2.6)

3. Primary Outcome: Trajectory Deviation
Description: Trajectory Deviation (TD) is assessed by comparing the actual motion trajectory with a predefined reference trajectory using the intelligent rehabilitation robot training system. TD is calculated as the mean Euclidean distance (in mm) between discrete points along the actual movement path and the nearest corresponding points on the reference trajectory. This metric provides a measure of point-specific accuracy and precision in following the ideal movement path, with smaller TD values indicating better trajectory control.
Time Frame: From enrollment to the end of treatment at 4 weeks
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | IRAT Group | RFE Group | CT Group
Number analyzed (Participants) | 25 | 26 | 25
millimeter
  baseline | 104.0 (7.9) | 100.7 (8.9) | 99.5 (8.3)
  4 weeks | 65.7 (8.0) | 98.1 (5.7) | 95.7 (4.7)

4. Primary Outcome: Trajectory Tracking Error
Description: Description:
  Trajectory Tracking Error (TTE) quantifies the cumulative deviation between the actual movement path and the predefined reference trajectory. It is computed as the sum of absolute differences in trajectory length between the two paths (in mm). TTE reflects overall movement efficiency and smoothness, capturing the patient's ability to maintain an optimal movement path throughout the task. A lower TTE indicates better movement planning and motor control.
Time Frame: From enrollment to the end of treatment at 4 weeks
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | IRAT Group | RFE Group | CT Group
Number analyzed (Participants) | 25 | 26 | 25
millimeter
  baseline | 60.8 (6.1) | 60.5 (6.0) | 61.6 (5.8)
  4 weeks | 36.8 (6.6) | 58.0 (2.8) | 59.1 (2.8)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | IRAT Group | RFE Group | CT Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The intervention period was relatively short and lacked long-term follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT06435624/Prot_SAP_000.pdf